CLINICAL TRIAL: NCT05338047
Title: Efficacy of Generic Pegfilgrastim vs Brand Name Pegfilgrastim for Neutrophil Recovery After Autologous Stem Cell Transplant
Brief Title: Efficacy of Generic Pegfilgrastim vs Brand Name Pegfilrastim for Neutrophil Recovery After Autotransplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Cesar Homero Gutierrez-Aguirre, Clinical Professor, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE22-00006
Record Dates: First submitted 2022-04-12; First posted 2022-04-20 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Myeloma Multiple; Lymphoma
Keywords: Autotransplant; Neutrophil recovery; Pegfilgrastim
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Generic pegfilgrastim (Placebo Comparator): One 6mg subcutaneous dose of generic pegfilgrastim in day+1 after autotransplant
  Interventions: Drug: Pegfilgrastim
- Brand name pegfilgrastim (Active Comparator): One 6mg subcutaneous dose of brand name pegfilgrastim in day+1 after autotransplant
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — Single 6mg dose of generic pegfilgrastim or brand name pegfilgrastim, at day +1 after autotransplant.
  Other Names: Neulasta; Linkix

SUMMARY:
This is a phase 2 clinical trial comparing time to neutrophil recovery after autotrasplant using generic pegfilgrastim vs brand-name pegfilgrastim.

DETAILED DESCRIPTION:
Thirty consecutive adults with lymphoma or myeloma receiving autologous peripheral blood stem cell transplant will be included in this phase 2 clinical trial. Patients will be allocated 1:1 in two groups: one subcutaneous 6 mg dose of generic pegfilgrastim (control group) or one 6mg dose of brand-name pegfilgrastim (intervention group) both at day +1 after the autotransplant. Daily complete blood counts were collected and time to neutrophil (>0.5x10^3/microL) and platelet recovery (>20x10^3/microL) will be obtained. The investigators will describe the proportion of adverse events and median time to neutrophil and platelet recoveries. Median or mean time to neutrophil recovery and time to platelet recovery will be calculated and compared with Mann-Whitney-Wilcoxon test or student T.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing autologous peripheral blood stem cell transplantation
* Patients with multiple myeloma or lymphoma
* Adults (>18 years)
* Both genders
* Eastern Cooperative Oncology Group (ECOG) <=2

Exclusion Criteria:

* Alanine Aminotransferase or bilirubin values >2.5 times the superior normal limit
* Creatinin >2.2mg/dL
* Fever >37.6°C
* Active infection
* Hepatitis B, C or HIV infection
* Congestive heart failure (ejection fraction <40%)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Time to neutrophil recovery | 15 days
  Time from autologous transplant to neutrophil count >0.5x10^3/microL

SECONDARY OUTCOMES:
Time to platelet recovery | 15 days
  Time from autologous transplant to platelet count >20x10^3/microL

CONTACTS AND LOCATIONS:
Overall Officials: Cesar H Gutierrez Aguirre, Principal Investigator — Hospital Universitario
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jagasia MH, Greer JP, Morgan DS, Mineishi S, Kassim AA, Ruffner KL, Chen H, Schuening FG. Pegfilgrastim after high-dose chemotherapy and autologous peripheral blood stem cell transplant: phase II study. Bone Marrow Transplant. 2005 Jun;35(12):1165-9. doi: 10.1038/sj.bmt.1704994. PMID 15880129
- [Result] Sheth V, Gore A, Jain R, Ghanekar A, Saikia T. Pegfilgrastim: More Cost Effective and Equally Efficacious Option as Compared to Filgrastim in Autologous Stem Cell Transplant. Indian J Hematol Blood Transfus. 2019 Jan;35(1):66-71. doi: 10.1007/s12288-018-0966-5. Epub 2018 May 17. PMID 30828150